CLINICAL TRIAL: NCT04384081
Title: A Phase I, Single-blinded, Randomized, Multiple Dose, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Different Dose Escalation Schemes of BI 456906 in Healthy Japanese Male Subject With BMI 23-40 kg/m2
Brief Title: A Study to Test How Different Doses of BI 456906 Are Tolerated in Japanese Men With a Body Mass Index (BMI) Between 23 and 40 kg/m2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1404-0021
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose group 1 (Experimental)
  Interventions: Drug: BI 456906
- Dose group 2 (Experimental)
  Interventions: Drug: BI 456906
- Dose group 3 (Experimental)
  Interventions: Drug: BI 456906
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 456906 — Solution for injection
  Arms: Dose group 1; Dose group 2; Dose group 3
Drug: Placebo — Solution for injection
  Arms: Placebo group

SUMMARY:
Main objectives are to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of different dose escalation schemes of BI 456906 in healthy Japanese male subject with BMI 23-40 kg/m2 and to determine a dose escalation scheme for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the assessment of the investigator, based on a complete medical history, a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests at screening visit
2. Japanese ethnicity, according to the following criteria:

   - born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
3. Age of 20 to 45 years (inclusive) at screening visit.
4. BMI of 23.0 to 40.0 kg/m2 (inclusive) with a minimum absolute body weight of 65 kg at screening visit and a stable body weight (defined as no more than 5% change) 3 months prior to screening visit.
5. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
6. Subjects who agree to minimize the risk of making their partner pregnant by fulfilling any of the following criteria starting from the first administration of trial medication until 90 days after last administration of trial medication

   * Use of adequate contraception, any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration.
   * Vasectomized (vasectomy at least 1 year prior to enrolment)
   * Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subjects female partner
7. HbA1c < 6.5% at screening visit

Exclusion Criteria:

1. Exposure to any glucagon-like peptide 1 receptor (GLP-1R) agonist (including combination products) within twelve months prior to screening visit, or any previous exposure to BI 456906, or history of relevant allergy or hypersensitivity (including allergy, intolerability or lack of efficacy to trial medication or drugs that belong to the GLP-1R agonist class)
2. Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned within 6 months after screening visit, e.g. hip replacement
3. Any evidence of a concomitant disease, baseline condition, or medical history assessed as clinically relevant by the investigator including:

   * Repeated measurement of supine blood pressure (BP) ≥160/95 mmHg, or pulse rate (PR) >90 bpm after 5 minutes of resting at screening visit.
   * Renal artery stenosis or evidence of labile blood pressure including symptomatic hypotension, or history of relevant orthostatic hypotension, fainting spells, or blackouts.
   * A marked baseline prolongation of Q wave to T wave (QT)/QTc (corrected) interval (such as QTc intervals that are greater than 450 ms at screening or an increase of 30 ms versus screening or any other relevant ECG finding at screening (e.g., type 2 second-degree atrioventricular (AV) block (Type Mobitz II) or third-degree AV block) and heart rhythm disturbances (e.g., bradycardia with baseline heart rate (HR) <45 bpm (in the absence of medications that lower the heart rate), or tachyarrhythmia or ventricular tachycardia).
   * Family history of long QT-syndrome, use of prescription or over-the-counter medications known to significantly prolong the QT or QTc interval at screening.
   * A history of pancreatitis or a history of/current increase of Amylase/Lipase > 1.5- fold Upper limit of normal (ULN)
   * Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening visit, except appropriately treated basal cell carcinoma of the skin, personal or family history of medullary thyroid carcinoma or history of multiple endocrine neoplasia syndrome type 2
   * Any clinical condition that requires continuous pharmacotherapy during the trial. Pharmacotherapy that potentially induce a change in body weight (for example anti-hyperglycemic, anti-depressant, diuretics, steroids, insulin, anti-psychotics) need to be stopped 6 months prior to screening visit
   * Cholecystectomy and/or prior surgery of the GI tract (including bariatric surgery) that could interfere with body weight or the pharmacokinetics (PK) of the trial medication or auxiliary medicinal products of the trial [paracetamol (acetaminophen)] except appendectomy and simple hernia repair.
   * Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
   * Chronic or relevant acute infections including viral hepatitis, human immunodeficiency virus (HIV) and/or syphilis.
   * History of relevant allergy or hypersensitivity (including allergy to trial medication or its excipients)
   * History of congestive heart failure New York Heart Association (NYHA) class IIIV or cardiovascular abnormalities such as ventricular or supraventricular arrhythmias. History of symptomatic ventricular tachycardia, or history of type 2 second-degree AV block (Type Mobitz II) or third-degree AV block.
   * Any of the following conditions or procedures within the last six months prior to screening: myocardial infarction, unstable angina, coronary artery bypass graft (e.g. carotid bypass, peripheral vascular diseases bypass), percutaneous coronary intervention (diagnostic angiograms are permitted), transient ischaemic attack, cerebrovascular accident (stroke) or decompensated congestive heart failure.
   * Any lifetime history of suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
   * Any suicidal ideation of type 2 to 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past 12 months (i.e. active suicidal thought without method, intent or plan; active suicidal thought with method but without intent or plan; active suicidal thought with method and intent but without specific plan; or active suicidal thought with method, intent and plan).
4. Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
5. Participation in another trial where an investigational drug has been administered within 60 days or 5 half-lives (whichever is longer) prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
6. Current smokers (defined as more than 10 cigarettes or 3 cigars or 3 pipes per day)
7. Inability to refrain from smoking on specified trial days
8. Alcohol abuse (consumption of more than 24 g per day) Further exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Cumulative percentage (%) of subjects withdrawn from up-titration by dose escalation scheme. | up to 113 days

SECONDARY OUTCOMES:
AUC0-168 (area under the concentration-time curve of BI 456906 in plasma over the time interval from 0 to 168h) | up to 113 days
Cmax (maximum measured concentration of BI 456906 in plasma) after first dose | up to 113 days

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://mystudywindow.com